CLINICAL TRIAL: NCT05296174
Title: Effects of Cognitive-Oriented Intervention on Perceived Social Support, Depression Symptoms, and Stress-coping Strategies in Patients With Major Depressive Disorder
Brief Title: Effects of Cognitive-Oriented Intervention on Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Collaborators: National Defense Medical Center, Taiwan (Other); Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, The Office of Research and Development, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TSGH-IRB -1-102-05-019
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Issue
Keywords: major depressive disorder; cognitive-oriented intervention
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive-oriented intervention program (Experimental): The intervention group received a 40 mins social support intervention program once a week lasting for 6 weeks.
  All participants were assessed by questionnaires before and after the intervention.
  Interventions: Other: cognitive-oriented intervention program
- received health education program (Active Comparator): The control group received health education activities with the same frequency as the intervention group.
  All participants were assessed by questionnaires before and after the intervention.
  Interventions: Other: health education activities program

INTERVENTIONS:
Other: cognitive-oriented intervention program — The experimental group was offered six 40-minute courses once a week.
  Arms: cognitive-oriented intervention program
Other: health education activities program — The control group was offered health education activities once a week.
  Arms: received health education program

SUMMARY:
The specific aims of the study were to explore the effects of the cognitive-oriented intervention program for promoting social support on perceived social supports, depression symptoms, and stress-coping strategies for patients with major depressive disorder in Taiwan.

DETAILED DESCRIPTION:
Background: Based on the 2010 World Health Organization declaration, depression will be ranked second among the global disease burden by 2020, second only to cardiovascular disease. It has become a disease that incurs high personal and social costs, and thus warrants considerable concern regarding its mitigation and early prevention.

Purpose: The specific aims of the study were to explore the effects of the cognitive-oriented intervention program for promoting social support on perceived social supports, depression symptoms, and stress-coping strategies for patients with major depressive disorder in Taiwan.

Method: This study adopted a randomized controlled trial (RCT). Patients with major depressive disorder were recruited from acute psychiatric wards in a medical center in Northern Taiwan. The study was conducted from July 1, 2015, to December 31, 2016; 105 patients met the inclusion criteria, and 100 patients agreed to participate in the study and completed the evaluation. The participants were randomly assigned to intervention group or control group. The intervention group received a 40 mins social support intervention program once a week lasting for 6 weeks, and the control group received health education activities with the same frequency as the intervention group. All participants were assessed by questionnaires before and after the intervention. Statistical analyses were performed by using descriptive statistics, independent sample t tests, and linear multiple regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with MDD by a psychiatrist
* over 20 years of age
* able to speak Mandarin or Taiwanese and able to write.

Exclusion Criteria:

* patients who were diagnosed with other psychiatric disorders
* with severe cognitive impairment or who could not make conversation acceptably were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
the Chinese Version of the Multidimensional Scale of Perceived Social Support (MSPSS) | before the intervention to 6 weeks (after the intervention)
  The MSPSS was developed by Zimet, Dahlem, Zimet and Farley (1988). It contains 12 questions, with four questions in each of three categories: (1) support from a significant other (significant other subscale); (2) support from family (family subscale); and (3) support from friends (friend subscale). This study adopts the Chinese version of the social support scale translated by Wang (2008). The higher the scale score meant the higher the perceived level of social support.
the Coping Orientations to Problems Experienced (COPE) inventory | before the intervention to 6 weeks (after the intervention)
  The is a four-point scale with a total of 60 questions, including 14 subscales, which include active coping, planning, and suppression of competing activities, restraint, and use of instrumental social support, and humor are tend to problem-focused coping. The higher the score, the more often the response strategy is adopted.
The Chinese version of the Beck Depression Inventory-II (BDI-II) | before the intervention to 6 weeks (after the intervention)
  The BDI-II has 21 questions. Higher scores indicated a greater degree of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Li Cheng, PhD, Principal Investigator — Department of Nursing, Mackay Medical College

IPD SHARING:
Plan to Share IPD: No